CLINICAL TRIAL: NCT06514781
Title: The Application of Different Sedation Protocols in ICU Patients With Severe Pneumonia
Acronym: ICU
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024020151
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Severe Pneumonia
Keywords: Severe pneumonia; Sedative
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Use cyclopofol group: Initially use propofol as the sedative medication, with a continuous usage duration of more than 48 hours.
- Control group: Initially use non-propofol sedative medications, with a continuous usage duration of more than 48 hours.

SUMMARY:
This study collected data from 600 patients with severe pneumonia to compare the duration of mechanical ventilation under different sedation regimens in real-world settings. It also evaluated and compared the sedation success rates, hemodynamic changes, and clinical outcomes of patients with severe pneumonia.

DETAILED DESCRIPTION:
The study subjects were patients with severe pneumonia hospitalized in the Department of Respiratory and Critical Care Medicine at Xiangya Hospital, Central South University, from January 2024 to December 2024. Patients meeting all the following criteria were enrolled: (1) diagnosed with severe pneumonia; (2) receiving mechanical ventilation and requiring sedation treatment; (3) age ≥ 18 years. Patients were excluded if they met any of the following conditions: (1) allergic to routine sedative or analgesic medications; (2) had not undergone pain and sedation assessment; (3) transferred to another hospital during treatment; (4) abandoned treatment and were discharged within <72 hours of treatment. Data on patient demographics, laboratory tests, chest imaging, respiratory support methods, severity of illness assessments, sedative medication usage, and clinical outcomes were collected. The duration of mechanical ventilation under different sedation regimens in real-world settings was compared, and the correlation between sedation success rates, hemodynamic changes, and clinical outcomes in patients with severe pneumonia was evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

(1)From February 1, 2023, to March 30, 2024, diagnosed with severe pneumonia in the Respiratory Intensive Care Unit of Xiangya Hospital, Central South University. The diagnosis of severe pneumonia is based on meeting at least one major criterion or three or more minor criteria:

1. Major criteria:

   ①Infectious shock requiring vasopressor therapy despite adequate fluid resuscitation;②Respiratory failure requiring tracheal intubation or mechanical ventilation.
2. Minor criteria:

   * Respiratory rate ≥ 30 breaths/min; ②Oxygenation index (PaO2/FiO2) ≤ 250;

     * Involvement of multiple lobes; ④Altered mental status and/or disorientation; ⑤Blood urea nitrogen ≥ 20 mg/dl (7.14 mmol/L); ⑥Systolic blood pressure < 90 mmHg requiring aggressive fluid resuscitation. (2)Patients receiving mechanical ventilation who require sedation treatment. (3)Age ≥ 18 years.

Exclusion Criteria:

1. Allergic to routine sedative or analgesic medications.
2. Patients who have not undergone pain and sedation assessment.
3. Patients transferred to another hospital during treatment.
4. Patients who abandon treatment and are discharged within less than 72 hours of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From February 1, 2023, to March 30, 2024, diagnosed with severe pneumonia in the Respiratory Intensive Care Unit of Xiangya Hospital, Central South University.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation duration | 2024.01-2024.12
  It is defined as the time from intubation (for patients intubated after ICU admission) or ICU admission (for patients already intubated upon ICU admission) to extubation

SECONDARY OUTCOMES:
The patient's sedation success rate | 2024.01-2024.12
  The level of sedation was assessed using the Richmond Agitation-Sedation Scale (RASS). Successful sedation was defined by meeting both of the following criteria: a) the proportion of time during the study medication period that the RASS score was between +1 and -2 was ≥ 70.0%; b) no rescue therapy was used.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan Li, Doctor, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China